CLINICAL TRIAL: NCT03295162
Title: Effects of Melatonin as a Novel Antioxidant and Free Radicals Scavenger in Neonatal Sepsis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mohamed Hussein Metwally (Other)
Responsible Party: Sponsor-Investigator, Mohamed Hussein Metwally, Assistant Lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pediatrics Dept-ASU
Record Dates: First submitted 2017-09-25; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sepsis A Group (Experimental): neonates diagnosed with Sepsis and will receive melatonin. 10 mg product as a total dose of 20 mg .together with conventional treatment of Neonatal sepsis
  Interventions: Drug: Melatonin 10 mg; Combination Product: Conventional treatment of neonatal sepsis
- Sepsis B Group (Sham Comparator): neonates diagnosed with Sepsis and willnot receive melatonin., they will recieve only the conventional treatment of Neonatal Sepsis
  Interventions: Combination Product: Conventional treatment of neonatal sepsis
- Control (No Intervention): healthy neonates, in whom sepsis will be ruled-out on the basis of absence of any clinical or laboratory evidence suggestive of infection.

INTERVENTIONS:
Drug: Melatonin 10 mg — Melatonin will be given at a total dose of 20 mg dissolved in 4 ml of distilled water via enteral route in two doses of 10 mg each(2 ml ), with a 1-hour interval. to one group together with conventional treatment
  Arms: Sepsis A Group
Combination Product: Conventional treatment of neonatal sepsis — Conventional treatment of neonatal sepsis including antibiotics,IV fluids, Total Parenteral Nutrition,etc...
  Arms: Sepsis A Group; Sepsis B Group

SUMMARY:
Assess the efficacy of melatonin as an adjuvant in the treatment of free radical disease in septic preterms receiving melatonin compared to those on conventional treatment through measuring the level of Malondialdehyde as a marker of oxidative stress and by comparing other clinical and laboratory parameters of sepsis in both groups.

DETAILED DESCRIPTION:
This is a randomized controlled trial. It will be provisionally conducted on 55 neonates admitted to the neonatal intensive care units (NICUs) of Ain Shams University Hospitals, Cairo, Egypt.

Inclusion criteria:

The study will include:Preterm infants (less than 37 weeks gestational age). Evidence of neonatal sepsis.

Exclusion Criteria: Neonate with evidence of any of the following will be excluded:

Infants with hypoxic ischemic encephalopathy. Infants on nothing per os. Infants with high oxygen needs either on invasive or non-invasive mechanical ventilation.

Group Classification:

Studied neonates will be completely evaluated and subsequently discriminated, into 2 main groups:Sepsis group: including neonates with proved sepsis. These will be subsequently randomized by permuted block randomization according to sequence of enrollment into:Subgroup A: neonates with odd numbers will receive melatonin.

Subgroup B: neonates with even numbers will not receive the medicine. Non Sepsis group: healthy neonates, in whom sepsis will be ruled-out on the basis of absence of any clinical or laboratory evidence suggestive of infection.

Diagnosis of neonatal sepsis will be established based on the presence of: risk factors of sepsis (e.g., prematurity, chorioamnionitis), any clinical evidence suggestive of sepsis, quantitative C-reactive protein (CRP) levels ≥6 mg/dL, Rodwell's hematological scores ≥3, with or without positive blood culture results

1. Comprehensive history taking including:

   A.Antenatal history: Maternal age, maternal diseases; Maternal diabetic control, maternal fever, infection, prolonged rupture of membranes >=18 hours, malodorous vaginal discharge.

   B.Natal history: Gestational age, sex, and mode of delivery. C.Postnatal history: APGAR score, Respiratory distress and/or cyanosis.
2. Gestational age will be estimated using the date of the last menstrual period, early antenatal ultrasound if present when available and confirmed by the new Ballard scoring system
3. Full clinical examination including: chest, cardiac, abdominal and neurological examination.
4. Clinical signs of infection: lethargy, irritability, prolonged capillary refill, tachycardia, respiratory distress, apnea, convulsions, abdominal distension, feeding intolerance, hyperglycemia, temperature instability and bleeding.
5. Assessment of the hemodynamic state of the neonates: mean arterial blood pressure (MABP), urinary output, temperature, capillary refill time.
6. Laboratory investigations Complete blood picture (CBC) with differential leucocytic count. C- reactive protein (CRP) quantitative assay. Blood cultures. MDA assay: blood samples will be collected in plain tubes from peripheral veins or central venous access. Samples will be allowed to clot before centrifugation for 15 minutes and serum will be stored at (-20 degree C) until MDA analysis using MDA competitive ELISA-kit.

   Blood samples will be collected from all included neonates at enrollment and in day one for healthy group.

   As for subgroup A, other samples will be withdrawn at 4 and 72 hours after melatonin administration to assess serum level of malondialdehyde while for subgroup B another sample will be withdrawn after 72 hours
7. Melatonin Medication:

   Melatonin 10 mg rapid release capsules (puritans pride) will be used. Melatonin will be given at a total dose of 20 mg dissolved in 4 ml of distilled water via enteral route in two doses of 10 mg each(2 ml ), with a 1-hour interval.(Gitto et al., 2000)
8. Treatment protocol: All neonates will be managed according to the protocol of NICU beside routine neonatal care.

Babies admitted to NICU will be bathed, placed in incubator, attached to monitor.

Cannula will be inserted, IV fluids is started and IV antibiotics. If there is respiratory distress: O2 or ventilation is started, usually feeds are delayed to day 2 or day 3 (or even later) according the severity of condition (clinical decision according to the attending neonatologist).

If no distress and the baby is well: trophic feeds will be started (10ml/kg/day milk), feeds are increased in 10-20ml/kg/day according to baby tolerance, and the condition of the baby (clinical decision according to the attending neonatologist), IV fluids are reduced gradually.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants ( less than 37 weeks gestational age). Evidence of neonatal sepsis

Exclusion Criteria:

Infants with hypoxic ischemic encephalopath Infants on nothing per os. Infants with high oxygen needs either on invasive or non-invasive mechanical ventilation.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Melatonin as an antioxidant and free radicals scavenger in Neonatal sepsis | 3 days
  efficacy of melatonin as an adjuvant in the treatment of free radical disease in septic preterms receiving melatonin compared to those on conventional treatment through measuring the level of Malondialdehyde as a marker of oxidative stress

SECONDARY OUTCOMES:
melatonin as an adjuvant in management of neonatal sepsis | 3 days
  efficacy of melatonin as an adjuvant in the treatment of septic preterms compared to those on conventional treatment and by comparing other clinical and laboratory parameters of sepsis in both groups

IPD SHARING:
Plan to Share IPD: Undecided